CLINICAL TRIAL: NCT05764096
Title: Executive Functioning and Sleep Fragmentation in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Istituto Universitario di Studi Superiori Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 2439
Record Dates: First submitted 2023-03-07; First posted 2023-03-10 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Healthy Volunteers
Keywords: COVID-19;executive functioning;quality of sleep
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients: 38 patients admitted to the intensive care unit due to COVID-19 contagion
  Interventions: Other: No intervention
- Healthy control participants: An age- and education-matched group of 38 healthy individuals who did not report a previous COVID-19 contagion
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This project aims to investigate executive functioning abilities (primary outcome) and quality of sleep (secondary outcome) in patients with COVID-19 (while distinguishing between those with and without sleep fragmentation), compared with an age- and education matched control group of healthy individuals who did not experience contagion. Prefrontal electrical activity will be recorded with EEG in patients, and related to sleep and cognitive-executive metrics.

The main questions it aims to answer are:

* is executive functioning impaired in COVID-19 patients compared with individuals who were not infected?
* is there a relationship between altered sleep and impaired executive functioning in COVID-19 patients?
* is such relationship related to altered prefrontal brain activitity in COVID-19 patients?

DETAILED DESCRIPTION:
While impaired executive functioning has been often reported in association with COVID-19 contagion, it is still unclear whether, and to what extent, executive deficits might be explained by an altered quality of sleep, that been also frequently reported in COVID-19 patients. On this basis, this project aims to investigate executive functioning abilities (primary outcome) in patients hospitalized for a COVID-19 contagion, while distinguishing between those with and without sleep fragmentation (quality of sleep; secondary outcome), compared with an age- and education matched control group of healthy individuals who did not experience contagion. To this purpose, 38 COVID-19 patients and 38 healthy controls will be administered questionnaires and cognitive tasks aimed to assess: a) executive functioning/inhibitory control (GoNogo task); b) quality of sleep (NOSAS; Insomnia Severity Index; Epworth sleepiness scale). Prefrontal electrical activity will be recorded with EEG in COVID-19 patients, and related to sleep and cognitive-executive metrics. Statistical analyses will be aimed to investigate: a) a possible decrease of executive skills in COVID-19 patients compared with healthy controls, and in COVID-19 patients with fragmented sleep compared with those with normal sleep; b) possible differences in the relationship between executive performance and quality of sleep across the three experimental groups; c) whether possible differences in such relationship relate to prefrontal brain activity in patients. The results of this study will provide novel insights into the consequences of COVID-19 at the cognitive level, thus informing about treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* For patients: current contagion from COVID-19
* For patients and controls:
* age>18 years
* absence of clinical conditions, cognitive and sensory deficits, and severe psychiatric disorders that would impair participation in research identified through clinical history.

Exclusion Criteria:

* current or past neuro-psychiatric disorder
* current or past sleep disorder

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 38 patients admitted to the intensive care unit due to COVID-19 contagion, plus an age- and education-matched group of 38 healthy individuals who did not report a previous COVID-19 contagion
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Executive/Inhibitory skills | Assessment day
  Performance in a GoNogo task

SECONDARY OUTCOMES:
Risk of sleep-disordered breathing | Assessment day
  NOSAS (Neck, Obesity, Snoring, Age, Sex)
Severity of nighttime and daytime components of insomnia | Assessment day
  Insomnia Severity Index
Sleepiness | Assessment day
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Ita, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Requests for sharing will assessed case by case, and data will be made available on reasonable request.